CLINICAL TRIAL: NCT02607111
Title: A New Anticoagulation Method Using Dalteparin in Quotidian and Nocturnal Home Hemodialysis Patients: A Prospective Study
Brief Title: A New Anticoagulation Method Using Dalteparin in Quotidian and Nocturnal Home Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 107283
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2016-09

CONDITIONS: Kidney Failure
Keywords: Dalteparin; Dosage; Home Hemodialysis
MeSH Terms: conditions — Renal Insufficiency | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Experimental): Dalteparin injected as a bolus into the arterial port of the hemodialysis machine every dialysis session for four weeks
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Drug: Dalteparin

SUMMARY:
This study evaluates the optimal dosage and safety of Dalteparin when used as an anticoagulant for hemodialysis therapies.

DETAILED DESCRIPTION:
Routine anticoagulation is required during hemodialysis treatments. In North America, the anticoagulant of choice for hemodialysis therapies is unfractionated heparin (UFH), whereas in Western Europe, it is low molecular weight heparin (LMWH). Dalteparin is more commonly used in Canada and has been approved for use in the in-centre thrice-weekly hemodialysis population at a fixed dose of 5000 units. However, there have been no published studies to assess the use of dalteparin in home quotidian and/or nocturnal hemodialysis therapies. Patients on frequent hemodialysis or nocturnal hemodialysis in the home will be converted to Dalteparin from Heparin for 4 weeks to evaluate the optimal dosage and to assess its safety in this population

ELIGIBILITY:
Inclusion Criteria:

* Currently undergoing short-hour daily and nocturnal hemodialysis through the home dialysis program at London Health Sciences Centre.

Exclusion Criteria:

* Patients with increased bleeding risks
* Currently on full dose anticoagulants
* Active bleeding
* Diabetic retinopathy
* Active cancer receiving treatment within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-08; Primary Completion 2018-07 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
The mean dalteparin dose for the daily home hemodialysis patients | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan Huang, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada